CLINICAL TRIAL: NCT02998255
Title: Effect of Single Dose of 2L PEG on Bowel Preparation in Average-risk Patients
Brief Title: Effect of Single Dose of 2L PEG on Bowel Preparation in Average-risk Patients Undergoing Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20162097-5
Record Dates: First submitted 2016-11-30; First posted 2016-12-20 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-07

CONDITIONS: Health Behavior
Keywords: PEG; Bowel preparation; Colonoscopy
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single dose of 2L PEG (Experimental): 2 L of PEG solution was used on the day of colonoscopy.
  Interventions: Drug: Single dose of 2L PEG
- Split-dose of 4L PEG (Active Comparator): Split-dose of 4l PEG was used before and on the day of colonoscopy
  Interventions: Drug: Split dose of 4L PEG

INTERVENTIONS:
Drug: Single dose of 2L PEG — Patients at average risk for inadequate BP were given instructions for bowel preparation through phone call a day before scheduled colonoscopy. Patients began to drink 2 L of PEG 4-6 hours before colonoscopy at a rate of 250 mL every 15 minutes.
  Arms: Single dose of 2L PEG
Drug: Split dose of 4L PEG — All patients at average risk for inadequate BP were given instructions for bowel preparation through phone call a day before scheduled colonoscopy. the participants began to drink the first 2 L of PEG at 7:00-9:00 PM on the day before colonoscopy at a rate of 250 mL every 15 minutes. On the day of the procedure, patients took the remaining 2 L 4-6 hours before colonoscopy.
  Arms: Split-dose of 4L PEG

SUMMARY:
Adequate quality of bowel preparation(BP) is important for colonoscopy. Several guidelines recommend that split-dose of 4L PEG should be used as a standard regime for BP. However, the high-volume PEG still results in lower compliance to the regime and increased cost.

Some high risk factors for inadequate BP have been identified, including old age, constipation, diabetes, the use of narcotics and prior history of inadequate BP. For average-risk patients without the high risk factors, the procedure of BP could be easier. In the previous study, with the use of single dose of 2L PEG, more than 90% of average-risk patients achieved adequate BP. Here investigators hypothesized that compared with the standard split dose of 4L PEG, single dose of 2L PEG may be not inferior in BP quality while may be accompanied with better tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colonoscopy;
* Patients with average risks for inadequate BP (Patients were identified average-risk if they did not meet any factor of the following risk factors):

  * Constipation
  * Diabetes
  * Parkinson's disease
  * History of stroke or spine cord injure
  * Prior history of inadequate bowel preparation
  * BMI>25
  * Use of tricyclic antidepressant or narcotics

Exclusion Criteria:

* History of colorectal resection;
* Suspected colonic stricture or perforation;
* Incomplete or complete bowel obstruction;
* Use of prokinetic agents or purgatives within 7 days;
* Toxic colitis or megacolon;
* Pregnancy or lactation;
* Unable to give informed consent;
* Haemodynamically unstable.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Actual)
Dates: Start 2016-12; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Rate of adequate bowel preparation(defined as a total BostonBowel Preparation Score ≥6 with each segmental BBPS≥2) | 1 year
  The adequacy of bowel preparation is defined as Boston Bowel Preparation Scale (BBPS), a 4-point scoring system applied to each of 3 broad regions of the colon: the right side, the transverse section, and the left side. They were summed to give the total BBPS score, which ranged from 0 to 9.The withdrawal procedure was recorded by vedios. The BBPS and segmental scores in each segment were judged by one endoscopist who was familiar with the criteria of BBPS and blinded to group allocation.

SECONDARY OUTCOMES:
Polyp detection rate | 1 year
Rate of adverse events | 1 year
  adverse events, such as vomiting, nausea, headache, abdominal pain
Cecal intubation rate | 1 year
Cecal intubation time | 1 year
Withdrawal time | 1 year
Willingness to repeat bowel preparation | 1 year
  The number of patients have a willingness to undergo a repeated bowel preparation if needed

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Department of gastroenterology, Qinghai Provincial People's Hospital, Xining, Qinghai
  - Department of gastroenterology, Shaanxi Second People's Hospital, Xi'an, Shaanxi
  - Endoscopic center, Xijing Hospital of Digestive Diseases, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No